CLINICAL TRIAL: NCT00300014
Title: Comparative,Randomized Study Between Intravitreal Triamcinolone Acetonide and Air-Fluid Exchange in Eyes With Post Vitrectomy Diabetic Vitreous Hemorrhage
Brief Title: Efficacy and Safety of Intravitreal Triamcinolone Acetonide in Eyes With Post Vitrectomy Diabetic Vitreous Hemorrhage
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Asan Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IVT in vitreous hemorrhage
Record Dates: First submitted 2006-03-07; First posted 2006-03-08 (Estimated); Last update posted 2007-06-13 (Estimated); Status verified 2007-06

CONDITIONS: Post Vitrectomy State; Recurrent Diabetic Vitreous Hemorrhage
Keywords: Post vitrectomy; Recurrent diabetic vitreous hemorrhage; Intravitreal triamcinolone injection

INTERVENTIONS:
Procedure: Intravitreal triamcinolone injection
Procedure: Air-fluid exchange

SUMMARY:
The Purpose of this study is compare the efficacy of intravitreal triamcinolone in clearing recurrent post-vitrectomy diabetic hemorrhage with conventional treatment, air-fluid exchange.

DETAILED DESCRIPTION:
Vitreous hemorrhage is the most common complication of vitrectomy for diabetic retinopathy. Despite measures to prevent and control this bleeding, it can lead to air-fluid exchange in the office or to additional surgery in the operating room. Air-fluid exchange does not result in clear vision immediately after the procedure, and the patient has to maintain a face-down position. Vitreous lavage, a more invasive procedure performed in the operating room, may give rise to complications such as iatrogenic retinal breaks, incarcerations of vitreous in the sclerotomy sites, retinal detachment, rubeosis iridis, neovascular glaucoma, infective endophthalmitis, and sympathetic ophthalmia. In contrast, IVT injection as a treatment of post vitrectomy diabetic vitreous hemorrhage is a less invasive procedure and provides more prompt visual recovery, while avoiding the face-down position.

We believe that the rapid clearing of vitreous hemorrhage results from as follows: (1) triamcinolone delivered in vitreous cavity can give rise to mechanical sediment entangled with remaining blood (2) direct vascular stabilizing effect may be induced (3) antiangiogenic effect may play a role.

ELIGIBILITY:
Inclusion Criteria:

* Previous vitrectomy due to proliferative diabetic retinopathy
* Recurrent diabetic vitreous hemorrhage

Exclusion Criteria:

* Monocular vision
* Uncontrollable intraocular pressure

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2006-01; Study Completion 2007-05

PRIMARY OUTCOMES:
day 1 : intraocular pressure, biomicroscope exam, fundus exam
day 7 : intraocular pressure, biomicroscope exam, fundus exam
2 weeks : intraocular pressure, biomicroscope exam, fundus exam
4weeks: intraocular pressure, biomicroscope exam, fundus exam, fluorescein angiography
2 months : intraocular pressure, biomicroscope exam, fundus exam
3months : intraocular pressure, biomicroscope exam, fundus exam
6 months : intraocular pressure, biomicroscope exam, fundus exam

CONTACTS AND LOCATIONS:
Overall Officials: Sun Young Lee, MD, Principal Investigator — Asan Medical Center; He Won Chung, MD, Principal Investigator — Asan Medical Center; Young Hee Yoon, MD, Principal Investigator — Asan Medical Center; June-Gone Kim, MD, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea